CLINICAL TRIAL: NCT03026296
Title: Healthy Life Centers - Municipal Health Care Service for Lifestyle Changes - a Multicenter Intervention Study on Changes Among Participants and Moderators for Changes Such as the Centers Capacity and Competence and the Participants Motivation
Brief Title: Healthy Life Centers - Municipal Health Care Service for Lifestyle Changes - a Multicenter Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Western Norway University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016/546-1
Record Dates: First submitted 2017-01-17; First posted 2017-01-20 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Musculoskeletal Disease; Obesity; Psychological Disorder
Keywords: Physical Fitness; Health Status; Exercise; Tobacco Use Cessation; Quality of Life; Healthy Diet; Health Promotion; Patient Education as Topic; Counseling
MeSH Terms: conditions — Musculoskeletal Diseases; Obesity; Mental Disorders; Motor Activity; Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participators in HLCs (Experimental): Adults with high risk of non-communicable diseases (musculoskeletal disease, obesity, physical distress) about to start a 3 months structural support for lifestyle change in a Healthy Life Center (HLC) in Norway
  Interventions: Behavioral: Healthy Life Center

INTERVENTIONS:
Behavioral: Healthy Life Center — Depending on what behavior participants aim to change, they get individual counselling using elements from motivational interviewing, group-based exercise twice a week, diet courses and tobacco secession courses during three months
  Other Names: Frisklivssentralen (Norwegian)

SUMMARY:
A Healthy Life Center (HLC, 'Frisklivssentrale') is a public community-based health service providing lifestyle support programs for physical activity, smoking cessation and diet, to inhabitants with increased risk for development of non-communicable diseases. HLCs intention is to reach physically inactive people who need guidance to get more physically active, and offer them a lifestyle program for three months or more.

The main aim of this study is to study whether the HLCs, organized according to the Norwegian Directorate of Health's guidelines for municipal healthy life centers, affects the participants short term (3 months) and long term (15 months) physical activity level. Also changes in diet, tobacco use, health related quality of life, physical fitness, anthropometry, self-efficacy, motivation, drug use, use of health services and work participation will be assessed. Secondary aim is to study whether there are any moderators, such as HLCs capacity, expertise, and collaboration with other services, that have significance for participants' change. Also it will be studied whether the HLCs result in larger changes in some subgroups (e.g. socioeconomic) of participants than in others.

ELIGIBILITY:
Inclusion Criteria:

* about to start structural support for lifestyle change (regarding physical activity, diet and/or tobacco cessation
* referred to a Healthy Life Center (HLC) from either primary physician, from other health care services or social services, or participants seeking contact themselves without a specific referral.

Exclusion Criteria:

* having participated in an HLC the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1022 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
physical activity | change from baseline to 3 months
  measured by accelerometer (ActiGraph GT3X+) for seven consecutive days
physical activity | change from 3 months to 15 months
  measured by accelerometer (ActiGraph GT3X+) for seven consecutive days

SECONDARY OUTCOMES:
Physical activity | change from baseline to 3 months
  assessed by questionnaire
Physical activity | change from 3 months to 15 months
  assessed by questionnaire
health related quality of life | change from baseline to 3 months
  assessed by SF-36 questionnaire
health related quality of life | change from 3 months to 15 months
  assessed by SF-36 questionnaire
Diet | change from baseline to 3 months
  assessed by questionnaire
Diet | change from 3 months to 15 months
  assessed by questionnaire
Tobacco use | change from baseline to 3 months
  assessed by questionnaire
Tobacco use | change from 3 months to 15 months
  assessed by questionnaire
Physical fitness | change from baseline to 3 months
  assessed by a standardized progressive walking protocol to a submaximal workload on a treadmill
Physical fitness | change from 3 months to 15 months
  assessed by a standardized progressive walking protocol to a submaximal workload on a treadmill
Body weight | change from baseline to 3 months
  measured on a scale digital weight
Body weight | change from 3 months to 15 months
  measured on a scale digital weight
Body Mass Index | change from baseline to 3 months
  body height measured by a Seca altimeter
Body Mass Index | change from 3 months to 15 months
  body height measured by a Seca altimeter
Waist circumference | change from baseline to 3 months
  measured by Seca measurement tape
Waist circumference | change from 3 months to 15 months
  measured by Seca measurement tape
Hip circumference | change from baseline to 3 months
  measured by Seca measurement tape
Hip circumference | change from 3 months to 15 months
  measured by Seca measurement tape

CONTACTS AND LOCATIONS:
Overall Officials: Riina Kiik, phd, Study Director — Norwegian University of Science and Technology; Erik Kyrkjebø, phd, Study Director — Western Norway University of Applied Sciences
Locations (4):
- Norway (4):
  - Frisklivssentrale, Drammen (plus 9 More Communities), Buskerud
  - Frisklivssentrale, Levanger (plus 4 More Communities), Nord-Trøndelag County
  - Frisklivssentrale, Bodo (plus 11 More Communities), Nordland County
  - Frisklivssentrale, Laerdal (plus 6 More Communities), Sogn Og Fjordane County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blom EE, Aadland E, Solbraa AK, Oldervoll LM. Healthy Life Centres: a 3-month behaviour change programme's impact on participants' physical activity levels, aerobic fitness and obesity: an observational study. BMJ Open. 2020 Sep 28;10(9):e035888. doi: 10.1136/bmjopen-2019-035888. PMID 32988939
- See also: Helsedirektoratet Frisklivssentraler — https://helsedirektoratet.no/folkehelse/frisklivssentraler